CLINICAL TRIAL: NCT04635605
Title: Evaluation of the Efficacy of Methylene Blue Administration in SARS-CoV2- Affected Patients: a Phase 2, Randomized, Placebo- Controlled, Single Blind Clinical Trial
Brief Title: Methylene Blue Treatment of COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Epatocentro Ticino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB treatment of COVID19
Record Dates: First submitted 2020-09-28; First posted 2020-11-19 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: SARS-CoV2
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Intervention Model Description: This is a phase 2 proof of concept, randomized, placebo controlled, single blind clinical trial on the efficacy of Methylene Blue against SARS-CoV-2 infection in patients with recently diagnosed SARS-CoV-2 infection
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylene Blue (Experimental): Methylene Blue 100 mg capsules. Patients will receive Methylene blue (MB) capsules of 100mg every 12 hours for a total of 5 days.
  Interventions: Drug: Methylene Blue
- control group (Active Comparator): The control intervention would be the group receiving 100 mg placebo capsules twice a day for five consecutive days
  Interventions: Drug: Control Test

INTERVENTIONS:
Drug: Methylene Blue — Treatment Group. Methylene Blue 100 mg capsules, twice a day for 5 consecutive days, will be added to the current therapy of the patient, if any.
  Arms: Methylene Blue
Drug: Control Test — Arm B: Control Group. Placebo capsules 100 mg twice a day for 5 consecutive days, will be added to the current therapy of the patient, if any.
  Arms: control group

SUMMARY:
Despite enormous progress in understanding COVID-19, there is little evidence that a solution, therapeutic or preventive, is close to being achieved. Repurposing of well known, widely available drugs represent an attractive approach to speed up availability of active treatments. Such substances as i.e. hydroxychloroquine and others, are already under investigation and in widespread off label use. For many reasons Methylene blue (MB), the oldest synthetic substance in medicine (1876 synthesized by BASF) is such a promising candidate for an active treatment against SARS-CoV-2 infected people and for COVID-19 patients.

ELIGIBILITY:
Inclusion criteria are:

* signed informed consent
* age ≥ 18 years
* microbiologically confirmed SARS-CoV-2 infection
* negative pregnancy test in women of child-bearing age

Exclusion criteria are:

* documented refusal to participate in the study
* known G-6-Phophatase deficiency
* treatment with a serotoninergic drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
to compare the viral load kinetics in the enrolled patients with a SARS-CoV-2 positive nasopharyngeal swab demonstrating a reduction of the area under the curve day 0- day 21 of at least 25% | day 0 - day 21
  As primary outcome we will measure the viral load kinetics in the enrolled patients. This means the viral load (expressed as cycled of replication with the PCR method and the number of RNA copies) at baseline and at each scheduled timepoint of the study

SECONDARY OUTCOMES:
To calculate the percentage of patients clearing SARS-CoV-2 by 3, 6, 9, 12, 15 and 21 days after diagnosis | 3, 6, 9, 12, 15 and 21 days after diagnosis
  We report the number of patients (expressed as percentage) with negative oro-pharyngeal swab at the scheduled time-points
To calculate the percentage of patients having a reduction of viral load of > 2 log by day 3 | day 3
  We calculate the number of patients (expressed as percentage) that have a decreased viral load (expressed as RNA copies) greater than 2 log by day three
To calculate the percentage of patients having a poor outcome as measured by the need of hospitalization for COVID-19 | 3, 6, 9, 12, 15, 21, 28 and 84 days after diagnosis
  We calculate the number of patients (expressed as percentage) that need hospitalization due to COVID-19, within the timeframe of the study
To calculate the percentage of patients alive | at 28-days and 84-days
  We calculate the number of patients (expressed as percentage) still alive at day 28 and 84 of samples collection
Safety and tolerability of the administered drug are registered as "adverse events", which are all symptoms related or supposed to be related to the drug that appeared after the drug intake and were NOT present at baseline or before | 3, 6, 9, 12, 15, 21, 28 and 84 days after diagnosis
  Safety and tolerability of the administered drug are registered as "adverse events", which are all symptoms related or supposed to be related to the drug that appeared after the drug intake and were NOT present at baseline or before Adverse events are expressed as present (1) or absent (0), in the dedicated data sheet which will be collected at each scheduled visit
To measure the compliance by calculating the number of capsules taken by the patient and the overall number of patients who complete the treatment | 3, 6, 9, 12, 15 and 21 days after diagnosis
  We calculate the number of pills (expressed as absolute number) taken by each enrolled patient during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Epatocentro Ticino, Lugano, Canton Ticino, Switzerland